CLINICAL TRIAL: NCT02356211
Title: Longitudinal Outcome in a Veterans Geriatric Multifactorial Falls Assessment Clinic: A Prospective Controlled Study
Brief Title: Longitudinal Outcome in a Veterans Geriatric Multifactorial Falls Assessment Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Powers, James S., M.D. (Individual)
Responsible Party: Principal Investigator, James S. Powers, MD, Associate Clinical Director, TVHS GRECC, Powers, James S., M.D.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 840
Record Dates: First submitted 2015-01-31; First posted 2015-02-05 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Aging
Keywords: falls

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Geriatric Multifactorial Falls Assessment Clinic
  Interventions: Other: Multifactorial Falls Assessment
- Control (No Intervention): Geriatric Evaluation and Management Service (GEM)

INTERVENTIONS:
Other: Multifactorial Falls Assessment — The Geriatric Multifactorial Falls Assessment Clinic is a component of GERIATRIC-PACT, a frail-elderly primary care patient-centered medical home with care provided by an inter-professional teamlet consisting of a geriatrician, geriatric nurse practitioner, clinical pharmacist, licensed practical nurse, nurse care manager, social worker, and dietitian. GERIATRIC-PACT operates with increased ancillary support compared to Primary Care PACT. Falls assessment patients were referred by primary care providers and were evaluated and treated by the GERIATRIC-PACT teamlet, including ordering of tests and medication adjustment, with an average of two visits and active follow-up for one year.
  Other Names: Falls Clinic
  Arms: Treatment

SUMMARY:
Objective To reduce subsequent falls following Multifactorial Falls Assessment Design: Prospective Case Control

Population: Frail elderly Veteran outpatient population referred for falls assessment

Methods: Prospective controlled trial of Geriatric Multifactorial Falls Assessment Clinic patients followed for 1 year and outcomes compared to Acute Geriatric Evaluation and Management (GEM) Inpatient Unit discharge control group.

DETAILED DESCRIPTION:
We designed a prospective controlled trial to compare the effectiveness of outpatient falls assessment and treatment for community-dwelling frail elderly patients with history of falls referred to an active management Geriatric Multifactorial Falls Assessment Clinic with a control group of patients discharged from an Acute Geriatric Evaluation and Management (GEM) Inpatient Unit during the same time period, but who were not specifically referred for falls assessment. We hypothesized that a population of frail elderly referred by their primary care physicians and who reported for evaluation to a Geriatric Multifactorial Falls Assessment Clinic would show a reduction in falls compared to controls, when provided a time-limited consult evaluation with active follow-up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling frail elderly with history of fall

Exclusion Criteria:

* Severe dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Powers, MD, Principal Investigator — TVHS GRECC
Locations (1):
- TVHS Nashville Campus, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Per Va IRB, no personal identifiers including age >89 can be shared. Aggregate data published: Powers JS, Samuels LR, Hu JR, Roumie CL. Veterans Geriatric Multifactorial Falls Assessment Clinic is Associated with Lower Fall Rate . J Gerontology and Aging Research 2017;1:102.

REFERENCES:
- [Result] Michael YL, Whitlock EP, Lin JS, Fu R, O'Connor EA, Gold R; US Preventive Services Task Force. Primary care-relevant interventions to prevent falling in older adults: a systematic evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2010 Dec 21;153(12):815-25. doi: 10.7326/0003-4819-153-12-201012210-00008. PMID 21173416
- [Result] Chang JT, Morton SC, Rubenstein LZ, Mojica WA, Maglione M, Suttorp MJ, Roth EA, Shekelle PG. Interventions for the prevention of falls in older adults: systematic review and meta-analysis of randomised clinical trials. BMJ. 2004 Mar 20;328(7441):680. doi: 10.1136/bmj.328.7441.680. PMID 15031239
- [Result] Moyer VA; U.S. Preventive Services Task Force. Prevention of falls in community-dwelling older adults: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2012 Aug 7;157(3):197-204. doi: 10.7326/0003-4819-157-3-201208070-00462. PMID 22868837
- [Result] Tinetti ME, Baker DI, McAvay G, Claus EB, Garrett P, Gottschalk M, Koch ML, Trainor K, Horwitz RI. A multifactorial intervention to reduce the risk of falling among elderly people living in the community. N Engl J Med. 1994 Sep 29;331(13):821-7. doi: 10.1056/NEJM199409293311301. PMID 8078528
- [Result] Panel on Prevention of Falls in Older Persons, American Geriatrics Society and British Geriatrics Society. Summary of the Updated American Geriatrics Society/British Geriatrics Society clinical practice guideline for prevention of falls in older persons. J Am Geriatr Soc. 2011 Jan;59(1):148-57. doi: 10.1111/j.1532-5415.2010.03234.x. PMID 21226685

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Geriatric Multifactorial Falls Assessment Clinic
  Multifactorial Falls Assessment: The Geriatric Multifactorial Falls Assessment Clinic is a component of GERIACTRIC-PACT, a frail-elderly primary care patient-centered medical home with care provided by an inter-professional teamlet consisting of a geriatrician, geriatric nurse practitioner, clinical pharmacist, licensed practical nurse, nurse care manager, social worker, and dietitian. GERIATRIC-PACT operates with increased ancillary support compared to Primary Care PACT. Falls assessment patients were referred by primary care providers and were evaluated and treated by the GERIATRIC-PACT teamlet, including ordering of tests and medication adjustment, with an average of two visits and active follow-up for one year.
- Control: Geriatric Evaluation and Management Service (GEM) The Geriatric Evaluation and Management Service (GEM) is an acute inpatient service with over 150 discharges annually. Frail elderly treated on GEM receive inter-professional geriatric team assessment and treatment while hospitalized. Patients discharged to home return to the care of their primary physicians.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 57 | 52
Completed | 54 | 42
Not Completed | 3 | 10
Not completed — Withdrawal by Subject | 2 | 2
Not completed — ineligible | 1 | 8

BASELINE CHARACTERISTICS:
Population: Intervention: 2 withdrawals, 1 bedfast, excluded from analysis Control: 2 withdrawals, 8 high functioning, excluded from analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 54 | 42 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 54 | 42 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.3 (8.8) | 74.1 (13.1) | 76.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 53 | 41 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 45 | 37 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 42 | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Falls
Description: Number of participants who experienced falls in 12 months, based on self-recall and telephone interview.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 55 | 51
Participants | 22 | 35

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Treatment: Geriatric Multifactorial Falls Assessment Clinic
  Multifactorial Falls Assessment: The Geriatric Multifactorial Falls Assessment Clinic is a component of GERIACTRIC-PACT, a frail-elderly primary care patient-centered medical home with care provided by an inter-professional teamlet consisting of a geriatrician, geriatric nurse practitioner, clinical pharmacist, licensed practical nurse, nurse care manager, social worker, and dietitian. GERIATRIC-PACT operates with increased ancillary support compared to Primary Care PACT. Falls assessment patients were referred by primary care providers and were evaluated and treated by the GERIATRIC-PACT teamlet, including ordering of tests and medication adjustment, with an average of two visits and active follow-up for one year. -- open label
- Control: Geriatric Evaluation and Management Service (GEM)
  The Geriatric Evaluation and Management Service (GEM) is an acute inpatient service with over 150 discharges annually. Frail elderly treated on GEM receive inter-professional geriatric team assessment and treatment while hospitalized. Patients discharged to home return to the care of their primary physicians.- open label
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 6/55 | 12/51
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/51
Other Adverse Events (participants affected / at risk) | 0/55 | 0/51

LIMITATIONS AND CAVEATS:
Fall rates determined by patient recall at 1 year by telephone interview. All patients were consented so advanced demented patients were not included in the intervention.

Falls e-consults were limited by EMR information and provider discretion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No